CLINICAL TRIAL: NCT05428267
Title: Sexual Dysfunction in Patients With Cirrhosis Before and After Liver Transplantation
Brief Title: Sexual Dysfunction in Cirrhosis
Acronym: SEDYC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP220052
Record Dates: First submitted 2022-06-10; First posted 2022-06-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Sexual Dysfunction in Patients With Cirrhosis Awaiting Liver Transplantation
Keywords: Cirrhosis; Sexual dysfunction
MeSH Terms: conditions — Fibrosis; Sexual Dysfunction, Physiological | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients on the liver transplant list for cirrhosis. (Experimental): Prevalence of sexual dysfunction before and after LT
  Interventions: Other: questionnaire; Other: blood collection

INTERVENTIONS:
Other: questionnaire — Completion of questionnaires (IIEF5/FSFI, SF 36, Fatigue Scale Score, Self Esteem Inventory, Hospital Anxiety and Depression Scale) during the pre-transplant consultation, then during a consultation 6 months after transplantation
Other: blood collection — Collection of 2 tubes of 5mL of blood during a scheduled blood draw in the patient's care pathway. This sample will also be taken after the transplant (6 months later)

SUMMARY:
The prevalence of erectile dysfunction (ED) is about 10% in the general population, but increases with age, ranging from 9.1% in men 40-49 years to 55% in men >70. The major risk factors for ED are as follows: diabetes; heart conditions; tobacco use; obesity; injuries to the nerves that control erection; medications such as antidepressants; psychological conditions such as stress, anxiety, or depression; and drug or alcohol use (4). The International Index of Erectile Function (IIEF5) is a simple and well-validated tool for the evaluation of ED (5) and is considered the gold standard for the diagnosis and evaluation of symptom severity. The link between cirrhosis and ED has been suggested in a recent study, showing ED was also impacted by liver failure, portal hypertension and other known risk factors. In the investigators team, they showed, additionally, that neurocognitive impairment is associated with ED in cirrhosis (data not published). The prevalence of ED after liver transplantation (LT) varies among series, ranging from 66 to 86%.

After LT, on the one hand, improvement of liver function and bioavailable testosterone favours the improvement of ED. On the other hand, immunosuppressive agents are suspected to worsen it.

ED's reversibility has also been discussed; nevertheless, data are scarce and heterogeneous.

In the investigators group, they can perform in routine a neurocognitive evaluation of patients with cirrhosis thanks to a neuropsychologist experienced in cognitive disorders occurring in patients with cirrhosis. The aims of this study are: 1) to compare the prevalence of erectile dysfunction (ED) in a population of patients with cirrhosis before liver transplantation (LT) and one year after LT; (2) to describe factors associated with ED before and after LT, with a special focus of hormonal profile, neurocognitive impairment, multimodal brain Magnetic resonance imaging (MRI) and of the type of immunosuppressive therapy used; (3) to assess the impact of ED on sexual partner; (4) to evaluate the efficacy of the treatment with phosphodiesterase-5 inhibitors (PDE-5) drugs after LT.

Methods: neurocognitive tests will be performed by an expert neuropsychologist. Biological evaluation will include an evaluation of liver function, hormonal assessment (bioavailable testosterone). MRI acquisition protocol will include anatomical sequences (3D-T1, FLAIR, T2, T2

*), diffusion tensor imaging (DTI) and two single voxel MR spectroscopy acquisitions. Evaluation will be performed before LT and 1 year after LT.

DETAILED DESCRIPTION:
PREVALENCE OF ERECTILE DYSFUNCTION IN PATIENTS WITH CIRRHOSIS BEFORE AND AFTER LIVER TRANSPLANTATION. EFFECTIVENESS OF PHOSPHODIESTERASE-5 INHIBITORS.

1. Research objectives The aims of investigators study are: (1) to compare the prevalence of erectile dysfunction (ED) in a population of patients with cirrhosis before liver transplantation (LT) and one year after LT; (2) to describe factors associated with ED before and after LT, with a special focus of hormonal profile, neurocognitive impairment, multimodal brain Magnetic resonance imaging (MRI) and of the type of immunosuppressive therapy used; (3) to assess the impact of ED on sexual partner; (4) to evaluate the efficacy of the treatment with phosphodiesterase-5 inhibitors (PDE-5) drugs before and after LT.
2. Scientific context (international + any preliminary results of the teams involved) Erectile dysfunction (ED) is defined as the inability to develop or maintain an erection during sexual intercourse (1, 2) and is the main concern in terms of sexual dysfunction among men. The prevalence of ED increases with age, ranging from 9.1% in men 40-49 years to 54.9% in men >70 years (3). The major risk factors for ED are as follows: diabetes; heart conditions; tobacco use; obesity; injuries to the nerves that control erection; medications such as antidepressants; psychological conditions such as stress, anxiety, or depression; and drug or alcohol use (4). The International Index of Erectile Function (IIEF5) is a simple and well-validated tool for the evaluation of ED (5) and is considered the gold standard for the diagnosis and evaluation of symptom severity. The link between liver diseases, especially cirrhosis, and ED has not been well established. Chronic liver disease, especially cirrhosis, may also be associated with an increased risk of ED (6,7). Hormonal abnormalities, such as hyperoestrogenism, are well-known consequences of liver failure. Data regarding the prevalence of ED are inhomogeneous, with reports varying from 63% to 93% (8, 9) in patients who are candidates for liver transplantation (LT). The largest study published to date in patients with cirrhosis (7) showed that ED in cirrhotic patients is impacted by liver function, portal hypertension and known risk factors, such as diabetes mellitus and arterial hypertension. More recently, a second study conducted in 102 patients with Child-Pugh A cirrhosis suggested that cirrhosis was not a risk factor for ED per se (10). Investigators recently conducted an observational monocentric study in patients with cirrhosis (manuscript under revision). Investigators confirmed that ED was very frequent in their population (85%). Investigators also found that the severity of liver disease, assessed by the MELD or Child-Pugh score, was an independent factor associated with ED. Moreover, investigators found a very strong correlation between neurocognitive performance, evaluated by the psychometric hepatic encephalopathy test score (PHES), and ED. Last, investigators observed that in the subgroup of patients with compensated cirrhosis, ED was significantly more frequent in patients with MHE than in patients without MHE. A recent brain MRI study has suggested that cortical volume and white matter microstructural changes were observed in patients with ED and showed significant correlations with clinical symptoms (11). The modifications of those features after treatment by PDE-5 have never been described. Data regarding the prevalence of ED after liver transplantation (LT) are heterogeneous and scarce. Two studies conducted in China (8, 9) have shown slight improvements in ED after LT. However, the results were obtained from a small cohort of patients, and the authors insisted on an association between post-LT ED and immunosuppressive therapy, which is an obvious confounding factor. In kidney transplantation, a recent meta-analysis has suggested that phosphodiesterase inhibitor drugs are efficient in ≈60%.
3. Implementation date and duration Investigators plan to implement the study in July 2019. Investigators aim to evaluate 100 patients before and one year after LT. As 110 LT are performed each year in investigator's centre (75% male gender), the study is going to last 2 years and a half.
4. Protocol

   • Type of study

   This is a prospective study that will be performed in La Pitié-Salpêtrière Hospital. For the purpose of this study, patients will be admitted in the investigator's team day hospital structure, where investigators routinely perform neurological and neuropsychological work-up of patients before LT, including neuropsychological assessment, biological sampling, multimodal MRI. This structure is completely automatized and requires nurses, a neuropsychologist, neurologists, and hepatologists in order to diagnose neurological disorders in hepatological situations. Patients' relatives also fill up questionnaires. All caregivers involved in patient's evaluation build a clinical conclusion at the end of the day hospital and give a detailed record to the patient.

   • Population

   All male patients referred to the investigator's team Hepatology Unit for an evaluation for LT will be proposed to participate to the study. Inclusion criteria are: (1) cirrhosis; (2) male gender; (3) non-urgent indication for LT. Exclusion criteria are: (1) clinical HE; (2) dementia; (3) language barrier; (4) past history of prostatic surgery.

   • Evaluation before LT

   Clinical evaluation Clinical examinations will be performed on the day of study enrolment. Liver function will be assessed using the Child-Pugh score and the Model for End-stage Liver Disease (MELD) score. Previous portal hypertension-related complications will be recorded, including HE, variceal bleeding, hepatocellular carcinoma, and ascites. Concomitant diseases will also be recorded, including hypertension, diabetes mellitus, hyperlipidaemia, metabolic syndrome, and previous history of ED. All medications will be recorded, especially beta-blockers, diuretics, benzodiazepines. Attention will be paid on past and present tobacco use.

   IIEF5 questionnaire The patients will be invited to complete the IIEF5 questionnaire (5). Briefly, 5 items are scored from 1 to 5 points for a minimum score of 5 and a maximum score of 25. ED is classified into the following categories: 5-10: severe ED; 11-15: mild ED; 16-20: moderate DE; and 21-25: no ED.

   Q1. Over the last month, how often were you able to get an erection during sexual activity? 0 No sexual activity 5 Almost always or always 4 Most times (much more than half the time) 3 Sometimes (about half the time) 2 A few times (much less than half the time) 1 Almost never or never

   Q2. Over the last month, when you had erections with sexual stimulation, how often were your erections hard enough for penetration? 0 No sexual activity 5 Almost always or always 4 Most times (much more than half the time) 3 Sometimes (about half the time) 2 A few times (much less than half the time) 1 Almost never or never

   Q3. Over the last month, when you attempted intercourse, how often were you able to penetrate your partner? 0 No sexual activity 5 Almost always or always 4 Most times (much more than half the time) 3 Sometimes (about half the time) 2 A few times (much less than half the time) 1 Almost never or never

   Q4. Over the last month, during sexual intercourse, how often were you able to maintain your erection after you had penetrated your partner? 0 No sexual activity 5 Almost always or always 4 Most times (much more than half the time) 3 Sometimes (about half the time) 2 A few times (much less than half the time) 1 Almost never or never

   Q5. Over the last month, during sexual intercourse, how difficult was it to maintain your erection to completion of intercourse? 0 No sexual activity 1 Extremely difficult 2 Very difficult 3 Difficult 4 Slightly difficult 5 Not difficult

   Neuropsychological evaluation The neuropsychologist will evaluate the presence of MHE. The psychometric HE test score (PHES) will be used to evaluate possible neuropsychological abnormalities. Briefly, the PHES is based on 5 tests: the digit symbol test (DST), the number connection test (NCT) parts A and B, the serial dot test (SDT), and the line tracing test (LTT). The results will be corrected for age and educational level and were analysed according to Spanish standards (http://www.redeh.org/phesapp/datosE.html). MHE was defined by a PHES equal to or less than - 4 (13). The Stroop EncephalApp will be evaluated in investigator's population. This very simple test (using smartphone) has been shown to have a good sensibility for the diagnosis of MHE in a multicenter US study (14). The psychophysical statuses of the patients will be assessed using the Self-Rating Anxiety Scale, the Self-Rating Depression Scale, the Brief Psychiatric Rating Scale, and a quality of life questionnaire (HRQOL questionnaire).

   Laboratory analysis Peripheral blood will be collected for routine blood tests and determination of liver function.

   Hormone analysis will be performed and will include testosterone, follicle-stimulating hormone (FSH), luteinising hormone (LH), prolactin, and sex hormone binding globulin.

   Assessment of ED on partner's sexual life The Index Sexual Life questionnaire is specifically designed to measure the impact of ED on female partner's sexuality (15). All partners will be proposed to fill it up on the day of patient's evaluation.

   Multimodal brain MRI The acquisition protocol will include anatomical sequences (3D-T1, FLAIR, T2, T2*), diffusion tensor imaging (to assess white matter injury) and MR spectroscopy (to evaluate MHE).

   • Management of ED before LT

   In the absence of contra-indication, a treatment with PDE-5 will be proposed to all patients diagnosed with ED. PDE-5 are routinely used for the treatment of ED; therefore there are no additional fees for patient's treatment. Efficacy of treatment will be evaluated 30 days after introduction of treatment by a single urologist who is currently seeing all patients with ED in investigator's unit. Data on safety, including hypotension, will also be recorded. Investigators chose not to use vardenafil, as a recent study suggested that this medication had no effect on portal pressure; among the PDE's-5 available, investigators will use tadalafil.
   * Evaluation after LT The same clinical, neurocognitive, biological, and MRI evaluation will be recorded one year after LT. As some patients will be treated with tadalafil before LT, investigators will first ask patients the real consumption of tadalafil after LT. Then investigators will evaluate ED after tadalafil withdrawal thanks to the IIEF5 questionnaire. Investigators will also detail the following items: length of hospitalisation after LT; date and number of urgent re-admissions after LT; type of immunosuppressive medication. Investigators will also evaluate the occurrence of de novo comorbidities after LT, such as hypertension, diabetes mellitus, and overweight.
   * Management of ED after LT AFEF In the absence of contra-indication, a treatment with PDE-5 will be proposed to all patients diagnosed with ED. Efficacy of treatment will be evaluated 30 days after introduction of treatment by a single urologist who is currently seeing all patients with ED in Investigator's unit.
   * Judgment criteria

   Primary outcome: to compare prevalence of ED before and after LT according to IIEF5. Secondary outcomes: (1) to evaluate factors associated with ED, including neurocognitive impairment, hormonal and psychological profil; (2) to assess the impact of ED on sexual partner; (3) to evaluate the efficacy of the treatment (PDE-5) drugs after LT.

   • Each person's involvement in research

   Selection, and clinical evaluation will be performed by investigators of the study (MR, FC). The nurses of the day hospital will perform biological analysis in routine. Neurocognitive evaluation will be performed by the same neuropsychologist (AS). MRI analysis will be performed by the same experienced neuroradiologist (DG). Data collection will be performed by one medical technical assistant (SC).
5. Methods of analysis of results including statistical analysis plan

Continuous variables will be reported as means±standard deviation (SD) or medians (95% CI), and categorical variables will be reported as numbers (n) and percentages. A Student's t test will be used for group comparisons of normally distributed data, and the Mann-Whitney U test to compare data without a normal distribution. Mac Nemar and Wilcoxon tests will be used for group comparisons between patients before and after LT. Multivariate binary logistic regression models will be used to determine the independent factors associated with the presence of ED after LT. Univariate analysis was performed first, and then all significant variables were entered into a multivariate model. NCSS statistical software (Kaysville, Utah USA) will be used for all statistical analyses.

5. Schedule Inclusions will begin in September 2019. End of inclusion: March 2021. Study completion: March 2022. 6. Funding justification

This is a total funding request. The day hospital organisation is already in place. Therefore, investigators will need for this study:

1. A neuropsychological evaluation (quarter time for 2 years 1/2= 25.000 euros)
2. A medical technical assistant for data collection (quarter time for 2 years 1/2=25.000 euros) 7. Expected benefits Investigators expect to assess: (1) the prevalence and (2) the factors mainly involved in ED in cirrhotic patients before and after LT (hormonal disturbance, neurological involvement, and drug toxicity). Secondly, investigators will be able to evaluate the efficacy of PDE-5 in patients with cirrhosis and in LT recipients. No data are available in the setting of LT. Investigators expect that prevalence of ED will be 85% before LT and 65% after LT. The likelihood of treatment efficacy should be 60% after LT. Therefore, investigators hope to observe a prevalence after treatment of 20%. Investigators do believe that a systematic screening of ED after LT and an adequate management could improve quality of life after LT.

ELIGIBILITY:
Inclusion Criteria:

* (1) cirrhosis; (2) non-urgent indication for LT.

Exclusion Criteria:

* (1) clinical HE; (2) dementia; (3) language barrier; (4) past history of prostatic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-07-26 (Estimated)

PRIMARY OUTCOMES:
Impact of liver transplantation on sexual dysfunction in patients with cirrhosis | through study completion, an average of 30 months
  The impact of liver transplantation on sexual dysfunction will be assessed by a comparison of questionnaires global results before and after the transplantation. For men investigators will use International Index of Erectile Function (IIEF5) questionnaire, and for women the Female Sexual Function Index (FSFI) questionnaire.

SECONDARY OUTCOMES:
Prevalence of sexual dysfunction in patients with cirrhosis. Safety issues No | through study completion, an average of 30 months
  This outcome will be assessed using IIEF5 questionnaire for men and FSFI questionnaire for women
Factors associated with sexual dysfunction in patients with cirrhosis | through study completion, an average of 30 months
  This outcome will be assessed using SF36 questionnaire
Hormonal concentration associated with sexual dysfunction in patients with cirrhosis | through study completion, an average of 30 months
  This result will be evaluated with biological statement carried out with the dosage of the following elements: FSH, LH, testosterone, sex-binding protein, dehydroepiandrosterone, dehydroepiandrosterone sulphate and androstenedione.
Prevalence of sexual dysfunction in patients who underwent liver transplantation | through study completion, an average of 30 months
  This outcome will be assessed using IIEF5 questionnaire for men and FSFI questionnaire for women

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'hépato-gastroentérologie Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided